CLINICAL TRIAL: NCT02066701
Title: Utility of Aberrant Gene Methylation in the Diagnosis of Barrett's Esophagus: Identification of Candidate Diagnostic Markers
Brief Title: Gene Methylation in the Diagnosis of Barrett's Esophagus: Identification of Candidate Diagnostic Markers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Other Study IDs: 12-001575
Record Dates: First submitted 2014-02-03; First posted 2014-02-19 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and cytology brushes will be stored for the duration of the study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endoscopy Barrett's: Patients undergoing clinically indicated upper endoscopy will be invited to participate. Patients who are known to have Barrett's Esophagus as well as patient who do not will be approached for enrollment
- Endoscopy control: Patients undergoing clinically indicated upper endoscopy will be invited to participate. Patients who are known to have Barrett's Esophagus as well as patient who do not will be approached for enrollment

SUMMARY:
This study is to identify potential markers from esophageal biopsies and brush cytology for feasibility of use in stool specimens for detection of Barretts Esophagus.

ELIGIBILITY:
Inclusion Criteria:

Controls: No endoscopic evidence of Barrett's Esophagus, able to give informed consent, 18 years of age or older.

Cases: At least 1 cm of visible columnar epithelium with intestinal metaplasia on histology confirmed by an expert GI pathologist (on biopsy), able to give informed consent, 18 years of age or older.

Exclusion criteria:

Controls: Patients with history of esophagectomy or mucosal ablation, gastrectomy, or known non-Barrett's esophageal pathology (e.g. eosinophilic esophagitis or achalasia), varices, esophagitis LA Grade B, C, D will be excluded. Patients with prior history of colon polyps or colon/esophageal/gastric/pancreatic carcinoma (unless had negative colonoscopy within 2 years to clear polyps).

Cases: Patients with history of esophagectomy or mucosal ablation, gastrectomy, or known non-Barrett's esophageal pathology (e.g. eosinophilic esophagitis or achalasia), will be excluded. Patients with prior history of colon polyps or colon/gastric/pancreatic carcinoma (unless had negative colonoscopy within 2 years to clear polyps).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for clinically indicated upper endoscopy will be approached to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
to determine if assay of aberrantly methylated gene markers can discriminate Barrett's Esophagus tissue (and presence of dysplasia) from esophageal squamous and gastric cardia tissue. | 1 day
  we will plan to identify the best markers from highly selected marker candidates to differentiate between subjects who have BE and those who do not have BE.

SECONDARY OUTCOMES:
Assess the accuracy of candidate markers in stool for detection of Barrett's Esophagus | One day
  Assess the ability of stool markers to distinguish between subjects who have BE and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States